CLINICAL TRIAL: NCT00123682
Title: Telephone Care Coordination to Improve Smoking Cessation Counseling
Brief Title: TeleQuit Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other); California Smokers' Helpline (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IMV 04-088
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Smoking
Keywords: Smoking Cessation; Care Management; Substance Use Disorder QUERI; Primary Care; Regional Expansion; Telephone
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 - proactive, intensive counseling (Experimental): Proactive outreach to counseling; multi-session counseling from California Smokers' Helpline
  Interventions: Procedure: Proactive outreach to counseling; Procedure: Intensive counseling
- Arm 2 - reactive, intensive counseling (Experimental): Reactive outreach to counseling; multi-session counseling from California Smokers' Helpline
  Interventions: Procedure: Reactive outreach to counseling; Procedure: Intensive counseling
- Arm 3 - proactive, self-help (Experimental): Proactive outreach to engage smoker in treatment; mailed self-help materials
  Interventions: Procedure: Proactive outreach to counseling; Procedure: Self-help
- Arm 4 - reactive, self-help (Experimental): Reactive approach to engaging smoker in treatment; mailed self-help materials
  Interventions: Procedure: Reactive outreach to counseling; Procedure: Self-help

INTERVENTIONS:
Procedure: Proactive outreach to counseling — Project staff reach out to engage referred smoker into telephone counseling
  Arms: Arm 1 - proactive, intensive counseling; Arm 3 - proactive, self-help
Procedure: Reactive outreach to counseling — Project staff send a letter to referred smoker, asking them to call to engage in telephone counseling
  Arms: Arm 2 - reactive, intensive counseling; Arm 4 - reactive, self-help
Procedure: Intensive counseling — Multi-session telephone counseling, delivered by California Smokers' Helpline
  Arms: Arm 1 - proactive, intensive counseling; Arm 2 - reactive, intensive counseling
Procedure: Self-help — Project staff send out self-help materials for smoking cessation
  Arms: Arm 3 - proactive, self-help; Arm 4 - reactive, self-help

SUMMARY:
TeleQuit is a group randomized trial testing whether a telephone care coordination program increases the rate of smoking cessation treatment for VA patients at study sites. We are testing whether proactive care coordination (counselor initiates the call to the patient) is more effective than reactive coordination (coordinator waits for the patient to call); and whether multi-session counseling is more effective than brief primary care-based counseling plus self-help materials. We randomly assigned study sites to either quitline counseling or brief counseling only. All patients receive brief smoking cessation counseling from their primary care physician, smoking cessation medications (once they are in contact with the VA care coordinator), and a follow-up call at 6 months. Care coordination will be provided by VA clinical staff. Intensive counseling is provided by the California Smokers' Helpline.

DETAILED DESCRIPTION:
Background:

Despite 40 years of progress, smoking remains the leading preventable cause of death in the United States, responsible for 435,000 deaths per year. Smoking is a particular problem within the VA, as VA users smoke substantially more than the general population across all categories of sex, age, and race. When adjusted for age and gender, the rate of smoking among VA users is 10% higher than the general US population - 33% vs. 23%. The prevalence of heavy tobacco users (defined as >20 cigarettes per day) in the VA is more than double that of the non-VA U.S. population (7.4% vs. 3.5%).

Current VA policy and new VA/DoD guidelines both mandate that patients be offered treatment (medications and counseling), regardless of whether they attend a smoking cessation program. Thus it is essential to treat patients within primary care, since most smokers interested in quitting cannot or will not attend a cessation program.

Objectives:

This project sought to make smoking cessation an area of excellence for two VA networks by adapting and expanding the primary care-based Telephone Care Coordination Program (TCCP) throughout Sierra Pacific Healthcare Network (VISN 21) and Greater Los Angeles Healthcare System (VISN 22).

This regional expansion built on the TCCP, a very successful VA Substance Use Disorder QUERI demonstration project implemented at two facilities. In the demonstration project, across the 10 intervention sites, there were 2,900 referrals for smoking cessation in 10 months. VA care coordinators proactively contacted patients and connected them with the California Smokers' Helpline. About 45% of patients starting treatment were abstinent six months later--equal to or better than smoking cessation clinics. A cost analysis showed substantial savings per quitter compared to provider-based and clinic-based programs.

Methods:

We developed a telephone-based smoking cessation program that was integrated as a routine clinical care option at five VISN 21 and VISN 22 facilities (38 clinic sites). Referrals to the program were generated by a provider during a visit through a brief consult in CPRS. Program staff then recruited patients and, after obtaining consent, enrolled the patients into treatment. Data were collected at the site level (quantity of referrals, service origins, etc.) and at the patient level (demographics, enrollment rates, abstinence rates at six months, etc.).

This project was a group randomized trial testing of whether telephone care coordination increases the rate of smoking cessation treatment. At the patient level, two questions are addressed:

1. Is proactive care coordination (counselor initiates the call to the patient) more effective than reactive coordination (coordinator waits for the patient to call)?
2. Is multi-session counseling more effective than brief primary care-based counseling plus self-help materials?

We randomly allocated all participating sites within VISNs 21 and 22 to either self-help or intensive counseling treatment arms. We randomly allocated each week of program referrals to either proactive or reactive care coordination. All patients received brief smoking cessation counseling from their primary care physician, smoking cessation medications (after study enrollment by the VA care coordinator), and a follow-up call at 6 months. Care coordination was provided by VA clinical staff (donated as in-kind support from the participating facilities). Intensive counseling was provided by the California Smokers' Helpline.

Status:

Complete except for ongoing data analysis.

ELIGIBILITY:
Inclusion Criteria:

* VA patient assigned to a clinic offering the program
* Smoker
* Patient wants to quit smoking

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3120 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Sherman, MD MPH, Principal Investigator — New York, NY
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, Sepulveda, California
  - New York, NY, New York, New York

REFERENCES:
- [Result] Fu SS, Sherman SE, Yano EM, van Ryn M, Lanto AB, Joseph AM. Ethnic disparities in the use of nicotine replacement therapy for smoking cessation in an equal access health care system. Am J Health Promot. 2005 Nov-Dec;20(2):108-16. doi: 10.4278/0890-1171-20.2.108. PMID 16295702
- [Result] Sherman SE, Takahashi N, Kalra P, Gifford E, Finney JW, Canfield J, Kelly JF, Joseph GJ, Kuschner W. Care coordination to increase referrals to smoking cessation telephone counseling: a demonstration project. Am J Manag Care. 2008 Mar;14(3):141-8. PMID 18333706
- [Derived] Sherman SE, Krebs P, York LS, Cummins SE, Kuschner W, Guvenc-Tuncturk S, Zhu SH. Telephone care co-ordination for tobacco cessation: randomised trials testing proactive versus reactive models. Tob Control. 2018 Jan;27(1):78-82. doi: 10.1136/tobaccocontrol-2016-053327. Epub 2017 Feb 11. PMID 28190003

RESULTS

PARTICIPANT FLOW:
Groups:
- Proactive Referral and Intensive Telephone Counseling: Proactive referral and intensive telephone counseling
- Reactive Referral and Intensive Counseling: Reactive referral and intensive counseling
- Proactive Referral and Self-help Materials: Proactive referral and self-help materials
- Reactive Referral and Self-help Materials: Reactive referral and self-help materials
Period: Overall Study
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials
Started | 1069 | 934 | 592 | 525
Completed | 749 | 731 | 438 | 430
Not Completed | 320 | 203 | 154 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials | Total
Number analyzed (Participants) | 1069 | 934 | 592 | 525 | 3120
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (10.8) | 54.2 (11.1) | 54.0 (11.8) | 55.1 (11.4) | 54.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 65 | 40 | 25 | 185
  Male | 1014 | 869 | 552 | 500 | 2935
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 5 | 3 | 5 | 26
  Asian | 31 | 16 | 19 | 8 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 231 | 200 | 73 | 71 | 575
  White | 605 | 543 | 342 | 289 | 1779
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 189 | 170 | 155 | 152 | 666
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 17.7 (9.9) | 18.3 (10.3) | 17.6 (10.2) | 20.1 (11.4) | 18.0 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Abstinence From Smoking
Time Frame: 6 month
Measure: Number; unit: percentage of participants
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials
Number analyzed (Participants) | 749 | 731 | 438 | 430
percentage of participants | 21 | 16.4 | 16.9 | 16.5

2. Secondary Outcome: Use of Cessation Medications
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials
Number analyzed (Participants) | 645 | 671 | 406 | 397
percentage of participants | 70.1 | 57.6 | 74.5 | 48.2

3. Secondary Outcome: Self-reported Quit Attempt
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials
Number analyzed (Participants) | 465 | 389 | 274 | 245
percentage of participants | 74 | 61.3 | 68.5 | 63

ADVERSE EVENTS:
Arm/Group | Proactive Referral and Intensive Telephone Counseling | Reactive Referral and Intensive Counseling | Proactive Referral and Self-help Materials | Reactive Referral and Self-help Materials
Serious Adverse Events (participants affected / at risk) | 0/1069 | 0/934 | 0/592 | 0/525
Other Adverse Events (participants affected / at risk) | 0/1069 | 0/934 | 0/592 | 0/525

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes